CLINICAL TRIAL: NCT07141745
Title: Electroporation vs. Radiofrequency Ablation Guided by 3D Imaging in Repeat Procedures for Atrial Fibrillation
Acronym: ERA-rePVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Stanisław Tubek, MD, PhD, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUBK.A460.25.068; SUBK.A460.25.068 (Other Grant/Funding Number: Wroclaw Medical University, Wroclaw, Poland)
Record Dates: First submitted 2025-07-31; First posted 2025-08-26 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation (AF); Ablation Techniques; Radiofrequency Catheter Ablation; Pulsed Field Ablation
Keywords: Atrial fibrillation re-ablation; Pulsed Field Ablation; Radiofrequency Catheter Ablation; Atrial firbillation reccurence
MeSH Terms: conditions — Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PFA group (Active Comparator): Patients in this arm will undergo 3D-mpping guided re-ablation with the PFA catheter
  Interventions: Procedure: Pulsed field ablation of reccurent atrial arrythmia
- RFA group (Active Comparator): Patients in this arm will undergo 3D-mpping guided re-ablation with RFA catheter
  Interventions: Procedure: Radiofrequency ablation of reccurent atrial arrythmia (standard of care)

INTERVENTIONS:
Procedure: Pulsed field ablation of reccurent atrial arrythmia — Substrate modification strategy based ablation of reccurent atrial arrythmia following pulmonary viens isolation employing pulsed field ablation with 3D guidance and high density mapping
  Arms: PFA group
Procedure: Radiofrequency ablation of reccurent atrial arrythmia (standard of care) — Standard radiofrequncy ablation of reccurent atrial arrythmia following pulmonary vien isolation employing substrate modification strategy
  Arms: RFA group

SUMMARY:
This is a prospective, randomized clinical trial evaluating the efficacy and safety of two techniques for repeat catheter ablation in patients with recurrent atrial fibrillation (AF): thermal energy ablation (radiofrequency) and non-thermal electroporation (pulsed field ablation), both guided by 3D imaging systems.

Patients undergoing repeat AF ablation will be randomly assigned to receive either thermal or electroporation ablation, performed according to standard hospital protocols. No additional invasive procedures are required. Following the ablation, participants will attend follow-up visits at 3, 6, and 12 months, including medical history review, physical examination, 12-lead ECG, and 24-hour Holter monitoring. Unscheduled ECG assessments will also be available if arrhythmia symptoms occur.

All study-related procedures are non-invasive and align with routine post-ablation care. Risks are limited to those typically associated with standard AF ablation procedures.

The main benefit of participation is close, structured follow-up by experienced electrophysiologists, allowing for early detection of arrhythmia recurrence and timely medical intervention when necessary.

Participant confidentiality and data protection will be ensured in accordance with GDPR regulations.

DETAILED DESCRIPTION:
Background Atrial fibrillation (AF) is one of the most common cardiac arrhythmias, with a lifetime risk of approximately 30% in individuals over 55 years of age. A primary treatment option for AF is pulmonary vein isolation (PVI), which targets the anatomical substrate of the arrhythmia. PVI can be achieved using thermal energy-either radiofrequency (RF) ablation or cryoablation-or with the newer, non-thermal method of pulsed field ablation (PFA). PFA delivers sequences of electrical pulses that cause selective electroporation of cardiomyocyte membranes, resulting in cell death while sparing adjacent non-cardiac tissues.

Despite these therapies, AF recurs in 30-50% of patients within the first year after ablation, regardless of the energy source used. The standard management for recurrence involves repeat ablation (re-PVI), targeting pulmonary vein reconnections and atrial substrate identified by electroanatomical mapping.

Randomized controlled trials comparing thermal modalities (RF vs. cryoablation) in first-time PVI have demonstrated similar safety and efficacy. Registry data and a single randomized trial suggest that PFA offers improved safety and comparable efficacy in initial PVI. However, no prospective randomized trial has evaluated the role of PFA in re-PVI.

Re-PVI procedures are technically more complex than index PVI, requiring high-resolution electroanatomical mapping of the left atrium to identify reconnection sites, followed by targeted ablation. While RF remains the established standard, growing evidence suggests that PFA may offer advantages due to its distinct mechanism of action, potentially overcoming thermal resistance from prior ablation. Retrospective data from our institution indicate that PFA may reduce procedure times and improve long-term success compared with RF, though these findings require confirmation in a controlled trial.

Study Overview This dual-center, prospective, randomized trial will compare the feasibility, safety, and efficacy of PFA versus RF ablation for re-PVI in patients with recurrent AF.

Study Design and Procedures Eligible patients admitted for clinically indicated repeat AF ablation at either the University Clinical Hospital in Wrocław (Department of Cardiology) or the University Clinical Hospital in Poznań (Department of Intensive Cardiac Therapy and Internal Medicine) will be invited to participate.

After providing informed consent, participants will be randomized in a 1:1 ratio to undergo either RF ablation or PFA. All procedures will include high-resolution electroanatomical mapping of the left atrium, followed by energy delivery according to the assigned modality. Post-ablation remapping will be performed to confirm acute procedural success.

Follow-up visits will take place at 3, 6, and 12 months, including medical history review, physical examination, 12-lead ECG, and 24-hour Holter monitoring. Additional visits and ECG assessments will be available if symptoms occur.

Data collected will include patient demographics, comorbidities, left atrial anatomy (by echocardiography), procedural characteristics (duration, fluoroscopy time, number and location of applications, acute isolation success, complications), and follow-up outcomes (late complications, arrhythmia recurrence, repeat ablation).

Study Locations Clinical Department of Cardiology, Jan Mikulicz-Radecki University Clinical Hospital, Wrocław, Poland Department of Intensive Cardiac Therapy and Internal Medicine, University Clinical Hospital, Poznań, Poland

Risks and Inconveniences Risks are consistent with standard AF ablation and are not increased by study participation. Potential complications include vascular access site events (bleeding, hematoma, arteriovenous fistula), stroke, or tamponade. No additional invasive procedures will be performed beyond routine ablation and follow-up. Participants must attend at least three scheduled outpatient visits.

Participant Characteristics Age: 18-85 years Gender: All Health status: Patients with AF recurrence after prior thermal PVI undergoing clinically indicated re-ablation Planned enrollment: Up to 250 participants

ELIGIBILITY:
Inclusion Criteria:

Documented recurrence of AF or atypical atrial flutter after prior PVI Eligibility for re-PVI

Exclusion Criteria:

Left ventricular ejection fraction < 30% Left atrial volume index (LAVI) > 72 mL/m² Untreated hyperthyroidism Hypertrophic cardiomyopathy Severe valvular heart disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial arrythmia in 12 month observation period | 12 months observation
  PFA is non-inferior to RFA in achieving freedom from documented atrial arrhythmia (AF, atrial flutter, or atrial tachycardia) lasting ≥30 seconds at 12 months after the index ablation procedure, as assessed by 12-lead ECG, 24-hour Holter monitoring, or symptomatic ECG recordings.

SECONDARY OUTCOMES:
Comparison of skin-to-skin time between PFA and RFA group | Data recorded during the procedure
  The parameter will be measured from vascular access to catheter removal.
Comparison of total fluoroscopy time between PFA and RFA group | Data recorded during the procedure
  The parameter is recorded by the electrophysiology system during the ablation procedure - total fluoroscopy exposure time (in seconds).
Comparison of total ablation time between PFA and RFA group | Data recorded during the procedure
  The parameter will be measured from the end of electroanatomical mapping to re-mapping.
Comparison of total radiation dose between PFA and RFA group | Data recorded during the procedure
  The parameter is recorded by the electrophysiology system during the ablation procedure as radiation dose (uGym2).
Safety endpoint | Adverse events during the index procedure and within following 90 days
  Occurrence of major adverse events within 90 days post-procedure, including but not limited to, cardiac tamponade, stroke or transient ischemic attack, pericardial effusion requiring intervention, pulmonary vein stenosis, atrioesophageal fistula, phrenic nerve injury, significant vascular access complications (e.g., bleeding requiring transfusion, pseudoaneurysm, arteriovenous fistula), symptomatic pulmonary vein stenosis

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Department of Cardio, Jan Mikulicz Radecki University Hospital in Wroclaw, Wroclaw, Poland